CLINICAL TRIAL: NCT07329998
Title: Oocyte Quality Assessment Using Spectrophotometer
Brief Title: The Aim of the Study is to Check Whether Follicular Fluid Evaluation Using a Spectrophotometer Can Differentiate High Quality Oocytes From Low Quality Oocytes. Oocyte Quality Will be Defined Using GDF9, BMP15 and Oocyte Morphology.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0069-23-HYMC
Record Dates: First submitted 2025-11-16; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Oocyte Quality Assessment Using Spectrophotometer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- follicular fluid evaluation using spectrophotometer to differentiate high low quality oocytes (Experimental)
  Interventions: Procedure: Oocyte quality assessment using spectrophotometer

INTERVENTIONS:
Procedure: Oocyte quality assessment using spectrophotometer — On the OPU (ovum pick-up) day the following blood biochemical markers will be measured as well- Blood interleukins 1-6, cytokine, hormone profile, lipid profile, cortisol.
  After collecting the oocytes- the Follicular fluid will be sent for the following tests-
  1. mid-infrared spectrometry,
  2. P, E2, testosterone, cortisol, cytokines, IL 1-6, lipids, fatty acids.
  3. BMP-15, GDF-9 and HSPG2
  4. GCMS-Gas Chromatography Mass Spectrophotometer

SUMMARY:
The aim of the study is to check whether follicular fluid evaluation using a spectrophotometer can differentiate high quality oocytes from low quality oocytes. Oocyte quality will be defined using GDF9, BMP15 and oocyte morphology. The correlation between cortisol levels in women and oocyte quality parameters will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-40 years.
* Undergoing IVF or IVF-ICSI treatment.
* At least five follicles visualized on ultrasound at the time of oocyte retrieval
* Ability to provide written informed consent.

Exclusion Criteria:

* Age >40 years.
* Fewer than five follicles at the time of oocyte retrieval.
* Use of donor oocytes.
* Significant medical comorbidities affecting ovarian function.
* Known ovarian malignancy or prior ovarian surgery significantly affecting follicular integrity.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-22 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Difference in follicular fluid infrared spectrophotometric profiles between high-quality and low-quality oocytes. | 3 Years
  Infrared spectrophotometric measurements of follicular fluid collected at oocyte retrieval will be obtained using attenuated total reflection Fourier-transform infrared spectroscopy (ATR-FTIR). Oocytes will be classified as high-quality or low-quality based on predefined morphological criteria and follicular fluid levels of GDF9 and BMP15 measured by ELISA. The primary outcome will be reported as differences in normalized spectral absorbance features between the two oocyte quality groups, including discrimination performance using multivariate analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel, Israel